CLINICAL TRIAL: NCT02206139
Title: Burn Out Among Surgical Residents Working at All Institutes in Lahore: An Area of Grave Concerns
Brief Title: Level of Burn Out of Surgical Residents Working in All Hospitals of Lahore
Status: Completed | Type: Observational
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Medical Officer, Services Hospital, Lahore
Other Study IDs: RBO102
Record Dates: First submitted 2014-07-24; First posted 2014-08-01 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Burn Out Syndrome
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The term burnout was coined by psychologist Herbert Freudenberger in 1974 in an article entitled "Staff Burnout" in which he discussed job dissatisfaction precipitated by work-related stress. A broadly applicable description defines burnout as a state of mental and physical exhaustion related to work or care giving activities. A long-standing conceptual and operational definition characterized burnout as a triad of emotional exhaustion (emotional over extension and exhaustion), depersonalization (negative, callous, and detached responses to others), and reduced personal accomplishment (feelings of competence and achievement in one's work) In the World Health Organization International Classification of Diseases, 10th revision, burnout is defined as a "state of vital exhaustion." Although no specific diagnosis of burnout is mentioned in the Diagnostic and Statistical Manual of Mental Disorders, burnout is a clear syndrome with significant consequences.

Burnout in health care professionals has gained significant attention over the last several years. Given the intense emotional demands of the work environment, clinicians are particularly susceptible to developing burnout above and beyond usual workplace stress. Residency training, in particular, can cause a significant degree of burnout, leading to interference with individuals' ability to establish rapport, sort through diagnostic dilemmas, and work though complex treatment decision making. Overall, burnout is associated with a variety of negative consequences including depression, risk of medical errors, and negative effects on patient safety. The goal of this review is to provide medical educators and leaders with an overview of the existing factors that contribute to burnout, the impact of burnout, inter specialty variation, and suggestions for interventions to decrease burnout.

ELIGIBILITY:
Inclusion Criteria:

* General Surgical resident

Exclusion Criteria:

* Residents of all other specialties
* All the General surgical consultants

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: General surgical residents of All the Hospitals Of Lahore
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
average working hours of residents | upto 3 months
  working hours of the residents will be noted and will be used this information to evaluate whether increased work hours lead to emotional instability and emotional exhaustion among them or not.

SECONDARY OUTCOMES:
emotional exhaustion | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sami Ullah, MBBS, Principal Investigator — SIMS/SHL
Locations (2):
- Pakistan (2):
  - Hospitals, Lahore, Punjab Province
  - Services Hospital Lahore, Lahore, Punjab Province